CLINICAL TRIAL: NCT05027464
Title: Developing and Testing a COVID-19 Vaccination Acceptance Intervention
Acronym: CoVAcS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency); Central Arkansas Veterans Healthcare System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SDR 21-141
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: COVID-19 Vaccination
Keywords: COVID-19 Vaccine; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: One-year cluster randomized parallel group trial, stratified by VISN, using covariate constrained randomization (e.g., rural/urban clinics, facility size). Specifically, the investigators will compare a Vaccine Acceptance Intervention versus Usual Care with randomization at the level of VA Medical Center (VAMC), with the intervention directed at VAMC clinic and CBOC PACT staff members.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study PIs and co-investigators, other research staff (except for the study statistician, see below), qualitative interviewers and participating VA staff will be unblinded because they are involved in delivering the intervention or, in the case of the qualitative researchers, will be tasked with interviewing study stakeholders about the intervention or implementation strategies. In contrast, the study evaluators, study statistician, and Veterans will be blinded to study arm assignment. Evaluators will conduct the study survey in Veterans, and while they will be aware of COVID-19 vaccination status, they will not be apprised of study arm. In addition, unless Veterans are unintentionally informed, Veterans will not know to which arm their VAMC has been randomized. Blinding of the study statistician conducting the outcomes analyses, survey evaluators, and the Veteran participants is important to protect the internal validity of study findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): The VAMC Internal Facilitator will partner with the trial External Facilitators (research team and designated External Facilitators in VISNS 16 and 21) to adapt and implement the study intervention to best meet the needs and preferences of their VAMC site. In addition, each CBOC and clinic affiliated with a VAMC in the Intervention arm will need to identify a Site Champion to provide clinic-specific information to facilitate implementation of the Vaccine Acceptance Intervention at their clinic or CBOC. In addition, for clinics and CBOCs assigned to the Vaccine Acceptance Intervention, VAMC, clinic and CBOC leadership will need to agree to release PACT staff for an initial two-hour Motivational Interviewing (MI) training, and at least one 60-minute post-training consultation session over the one-year trial period. There will be additional consultation sessions offered to intervention clinics and CBOC staff, but these will be optional.
  Interventions: Behavioral: Moving to COVID-19 Vaccine Acceptance Intervention
- Usual Care Arm (No Intervention): A VAMC assigned to Usual Care will have no specific trial intervention requirements beyond their usual level of participation in national and local initiatives to improve COVID-19 vaccine acceptance. At both Intervention and Usual Care sites, the study team will perform quarterly "environmental scans". The environmental scan survey will include questions about site specific barriers to COVID-19 vaccination (first dose and second dose if needed), current programs/initiatives in the clinic or local community that are improving or have had no impact on vaccination rates, and the perceived importance that the VAMC/CBOC clinic staff is placing on vaccination (Environmental Scan Survey, in preparation). At Usual Care sites, a point of contact will be chosen from each clinic and CBOC to complete the environmental scan, and at Intervention sites, the Site Champion (see below) will perform the quarterly scan.

INTERVENTIONS:
Behavioral: Moving to COVID-19 Vaccine Acceptance Intervention — The intervention utilizes a multi-pronged approach to increase Veteran vaccine acceptance. First, the research team will train Health Behavior Coordinators (HBCs) at VAI sites. HBCs will then train PACT teams at their site and Whole Health Coaches, Peer Specialists and other VA Staff in VAI strategies to use with unvaccinated Veterans. Whole Health Coaches, Peer Specialists and other VA Staff will conduct outreach calls, using strategies, with unvaccinated Veterans.
  Arms: Intervention Arm

SUMMARY:
The COVID-19 pandemic has resulted in significant loss of life and suffering with total case and death counts increasing daily, particularly with the emergence of the delta variant. COVID-19 vaccines have proven highly effective in preventing severe illness, hospitalization, and death. Nevertheless, according to VA data sources, only 56% of all U.S. Veterans have been vaccinated to date, largely owing to vaccine hesitancy and lack of access to vaccination. Thus, there is a critical need for evidence-based interventions to increase COVID-19 vaccine acceptance and access among Veterans, many of whom are vulnerable to poor outcomes of COVID-19. The overall goal of this study is to increase COVID-19 vaccination in Veterans of VISNs 16 and 21 who remain unvaccinated either because of vaccine hesitancy or lack of access to COVID-19 vaccine. Specifically, the investigators will test a COVID-19 Vaccine Acceptance Intervention (Motivational Interviewing) plus Implementation Facilitation.

DETAILED DESCRIPTION:
For Aim 1, the investigators will conduct a one-year cluster randomized controlled trial of a Vaccine Acceptance Intervention versus Usual Care with randomization at the level of VA Medical Center (VAMC). Usual Care will consist of all national and local initiatives to promote COVID-19 vaccine acceptance in Veterans such as vaccine mandates, mobile clinics, outreach calls, etc. The Implementation Facilitation team will include a VISN-level external facilitator, VAMC-level internal facilitators, and clinic-level site champions to support PACT staff, Coaches and Peers in implementing the Vaccine Acceptance Intervention with unvaccinated Veterans as well as in lowering barriers to vaccine access at intervention sites. For Aim 2, the investigators will identify a diverse sample of 450 Veterans across VAMCs in VISNs 16 and 21, who have had primary care visits at Intervention and Usual Care sites, and who have either recently received (N=360) or have not received (N=90) COVID-19 vaccination. The investigators will over sample recently vaccinated Veterans to describe the impact of the Vaccine Acceptance Intervention on Veterans' decisions to accept COVID-19 vaccination in addition to over-sampling women, ethnic/racial minorities, rural and younger Veterans, and those with mental health conditions. Follow-up qualitative interviews will be conducted in a subsample to better understand factors related to recent vaccine acceptance and persistent vaccine hesitancy. Finally, for Aim 3, the investigators will conduct process and summative interviews with VA staff and providers from VAMC sites in VISNs 16 and 21 with high and low vaccination rates) to learn which implementation strategies were most and least effective.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria by Aim:

* Aim 1: Primary care clinic visit in VISN 16 or 21
* Aim 2: =1 visit(s) at a participating VISN 16 or 21 primary care clinic or CBOC after the start of the trial at their site, and at the time of recruitment, COVID-19 vaccination status is verified as one of the following:

  * has not initiated COVID-19 vaccination
  * has initiated one of the two mRNA vaccines and is outside the window for the second dose
  * recently completed COVID-19 vaccination (has completed two doses of mRNA vaccination or has completed the single-dose Janssen/Johnson & Johnson vaccine within the past 60 days)
* Aim 3: Implementation-focused Interviews with VISN 16 and 21 Staff and HCPs

Exclusion Criteria:

Exclusion Criteria by Aim:

* Aim 1: Per VISN or VAMC leadership, the clinic or CBOC has extreme staffing shortages such that it would not be feasible or in the best interests of patient care to allow clinic or CBOC staff release time to participate in trainings or other meetings related to the trial
* Aim 2: Has initiated COVID-19 vaccination with one of the mRNA vaccines and is within the window to complete the second dose on schedule (< 42 days since dose 1)

  * Serious allergic reaction or other contraindication to COVID-19 vaccination or other vaccines (e.g., flu vaccine)
  * Currently in hospice care or < 6 months to live
  * No consistent ability to be contacted by phone
  * Participating in another COVID-19 trial or study (research study flag)
  * Moderate to severe dementia as documented in the patient's VA medical record
  * Increased suicide risk as indicated by behavioral health flag
* Aim 3: Staff or HCPs declines invitation to participate in the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338718 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Seal, MD MPH, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA; Jeffrey M Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR; Jennifer K Manuel, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pyne JM, Seal KH, Manuel JK, DeRonne B, Oliver KA, Bertenthal D, Esserman D, Purcell N, Petrakis BA, Elwy AR. Developing and testing a COVID-19 vaccination acceptance intervention: A pragmatic trial comparing vaccine acceptance intervention vs usual care - Rationale, methods, and implementation. Contemp Clin Trials. 2023 Oct;133:107325. doi: 10.1016/j.cct.2023.107325. Epub 2023 Aug 29. PMID 37652356
- [Result] Seal KH, Bertenthal D, Manuel JK, Pyne JM. Association of Demographic, Clinical, and Social Determinants of Health With COVID-19 Vaccination Booster Dose Completion Among US Veterans. JAMA Netw Open. 2022 Jul 1;5(7):e2222635. doi: 10.1001/jamanetworkopen.2022.22635. PMID 35852805

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: VAHCS
Groups:
- Intervention Arm: The VAHCS Internal Facilitator will partner with the trial External Facilitators (research team and designated External Facilitators in VISNS 16 and 21) to adapt and implement the study intervention to best meet the needs and preferences of their VAHCS site. In addition, each CBOC and clinic affiliated with a VAHCS in the Intervention arm will need to identify a Site Champion to provide clinic-specific information to facilitate implementation of the Vaccine Acceptance Intervention at their clinic or CBOC. In addition, for clinics and CBOCs assigned to the Vaccine Acceptance Intervention, VAHCS, clinic and CBOC leadership will need to agree to release PACT staff for an initial two-hour Motivational Interviewing (MI) training, and at least one 60-minute post-training consultation session over the one-year trial period. There will be additional consultation sessions offered to intervention clinics and CBOC staff, but these will be optional.
  Moving to COVID-19 Vaccine Acceptance Intervention: The intervention utilizes a multi-pronged approach to increase Veteran vaccine acceptance. First, the research team will train Health Behavior Coordinators (HBCs) at VAI sites. HBCs will then train PACT teams at their site and Whole Health Coaches, Peer Specialists and other VA Staff in VAI strategies to use with unvaccinated Veterans. Whole Health Coaches, Peer Specialists and other VA Staff will conduct outreach calls, using strategies, with unvaccinated Veterans.
- Usual Care Arm: A VAHCS assigned to Usual Care will have no specific trial intervention requirements beyond their usual level of participation in national and local initiatives to improve COVID-19 vaccine acceptance. At both Intervention and Usual Care sites, the study team will perform quarterly "environmental scans". The environmental scan survey will include questions about site specific barriers to COVID-19 vaccination (first dose and second dose if needed), current programs/initiatives in the clinic or local community that are improving or have had no impact on vaccination rates, and the perceived importance that the VAMC/CBOC clinic staff is placing on vaccination (Environmental Scan Survey, in preparation). At Usual Care sites, a point of contact will be chosen from each clinic and CBOC to complete the environmental scan, and at Intervention sites, the Site Champion (see below) will perform the quarterly scan.
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care Arm
Started (In this cluster randomized trial, VAHCS sites are randomized to the intervention arm where providers employed by facilities associated with the VAHCS, however outcomes are measured on the Veteran-level where Veterans are seen by providers.) | 148291; 5 VAHCS | 190427; 5 VAHCS
Completed | 148291; 5 VAHCS | 190427; 5 VAHCS
Not Completed | 0; 0 VAHCS | 0; 0 VAHCS

BASELINE CHARACTERISTICS:
Population: Veterans who had at least one primary care visit during the study period
Units Other Than Participants: VAHCS
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 148291 | 190427 | 338718
Number analyzed (VAHCS) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (15.1) | 62.9 (16.0) | 63.1 (15.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14406 | 18094 | 32500
  Male | 131215 | 168777 | 299992
  Unknown | 2670 | 3556 | 6226
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 84404 | 130970 | 215374
  Race: Black or African American | 32918 | 32313 | 65231
  Race: Asian | 8451 | 3918 | 12369
  Race: Native Hawaiian or Other Pacific Islander | 6192 | 2050 | 8242
  Race: American Indian or Alaska Native | 1081 | 1810 | 2891
  Race: Unknown | 15245 | 19366 | 34611
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 129305 | 161567 | 290872
  Ethnicity: Hispanic or Latino | 9005 | 17336 | 26341
  Ethnicity: Declined to Answer | 1717 | 2655 | 4372
  Ethnicity: Unknown | 8264 | 8869 | 17133
Region of Enrollment [Number; unit: participants]
  United States | 148291 | 190427 | 338718
Baseline Primary Series Rate (Randomization Unit Level) [Mean (Standard Deviation); unit: Percent of Participants] — This baseline measure was the percent of the randomization unit's participants that completed the COVID-19 vaccine primary series at the time of randomization and was used during covariate-constrained randomization to balance study arms by higher and lower vaccination rates. Population: The number of units for this baseline measure are the number of randomization units assigned to each arm (i.e., 5 and 5). This measure is percentage of participants in each randomization unit who completed primary series at the time of randomization
  Percent of Participants | 61.8 (6.30) | 64.2 (6.60) | 63.0 (5.89)
Marriage Status [Count of Participants; unit: Participants]
  Divorced/Separated | 38165 | 49476 | 87641
  Married/Common Law | 80240 | 105951 | 186191
  Single/Never Married | 22233 | 25002 | 47235
  Unknown | 2786 | 2514 | 5300
  Widow/Widower | 4867 | 7484 | 12351
Rurality [Count of Participants; unit: Participants]
  Highly Rural | 1399 | 1514 | 2913
  Rural | 40958 | 59849 | 100807
  Unknown | 2709 | 28 | 2737
  Urban | 103225 | 129036 | 232261
Care Assessment Needs (CAN) Score 1 Year Event Probability [Mean (Standard Deviation); unit: Probability] — The CAN score is a comorbidity index defined as a probability of being hospitalized or of mortality within a year. The CAN score was determined at baseline in this study and is used as a covariate in primary analyses.
  Probability | 0.181 (0.175) | 0.179 (0.174) | 0.180 (0.174)

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Any Dose COVID-19 Vaccination
Description: A greater proportion of Veterans in the intervention group will receive any dose of COVID-19 vaccination compared to usual care.
Time Frame: 1 year
Population: Veterans with at least one primary care visit during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 148291 | 190427
Participants | 57621 | 65407
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; Generalized linear mixed model to account for patient demographics and hierarchical levels for clinics nested within VAHCS. Null hypothesis is that both arms perform equivalently in vaccine uptake after a year. Power was based on recruited VAHCSs and at least 1,000 Veterans per clinic. Using two-sided 0.05 type I error rate, 5-20% outcome rate in UC, we have 90% power to detect between a 9.6% and 14.6% difference with a total sample size of 90,000 to 100,000; Test type: Superiority; p = 0.202, Regression, Logistic — Not adjusted for multiple comparisons; a priori threshold was P < 0.05; Patient demographics were fixed effects, and randomization units with clinics nested within randomization units were random effects; Odds Ratio (OR) = 1.249, 95% CI 2-sided [0.888 to 1.759] — An odds ratio above one indicates favoring the intervention arm over the usual care arm
Statistical Analysis 2: Comparison: Intervention Arm vs Usual Care Arm; Sensitivity analysis, same null hypothesis and model as primary analysis but different pool of patients: Not constrained to Veterans with at least one primary care visit; Test type: Superiority; p = 0.247, Regression, Logistic; Odds Ratio (OR) = 1.228, 95% CI 2-sided [0.867 to 1.738]
Statistical Analysis 3: Comparison: Intervention Arm vs Usual Care Arm; Sensitivity analysis; same model and null hypothesis but reassigning small clinics to their parent VAHCS facility, small meaning < 100 participants. This data set uses the primary analysis data set with the primary visit constraint; Test type: Superiority; p = 0.455, Regression, Logistic; Odds Ratio (OR) = 1.263, 95% CI 2-sided [0.684 to 2.334]
Statistical Analysis 4: Comparison: Intervention Arm vs Usual Care Arm; Sensitivity Analysis: same model and null hypothesis as primary outcome but the source of vaccination records omits Medicare claims data. The primary data source had included Medicare claims data on vaccination records as a supplement to the VA data; Test type: Superiority; p = 0.364, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.765 to 2.075]
Statistical Analysis 5: Comparison: Intervention Arm vs Usual Care Arm; Sensitivity Analysis: same model and null hypothesis as primary analysis model but the source of data is supplemented by state level registries, named "IZ Gateway", which was deployed summer of 2023 where Veteran records of vaccination could be updated at the VA from external vaccination facilities if the Veteran entered the VA in the same state as that vaccination facility. The primary analysis data contains Medicare claims data in this analysis, too; Test type: Superiority; p = 0.168, Regression, Logistic; Odds Ratio (OR) = 1.268, 95% CI 2-sided [0.904 to 1.778]

2. Secondary Outcome: Primary Series Completion of COVID-19 Vaccination
Description: A greater proportion of previously unvaccinated Veterans in the intervention arm will complete the primary series for COVID-19 vaccination compared to usual care
Time Frame: 1 year
Population: Veterans without any COVID-19 vaccination prior to study start who also had at least one primary care visit during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 29904 | 43939
Participants | 378 | 533
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; Power calculation is similar to the calculation for the primary outcome. Null hypothesis is described in the outcome comparison related to this statistical analysis plan; Test type: Superiority; p = .976, Regression, Logistic — P < 0.05 and no multiple comparison adjustment; We adjusted for patient demographics as fixed effects and randomization units and associated clinics as a three-level random effect; Odds Ratio (OR) = 0.993, 95% CI 2-sided [0.643 to 1.535] — An odds ratio above one indicates favoring the intervention arm over the usual care arm
Statistical Analysis 2: Comparison: Intervention Arm vs Usual Care Arm; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.893, Regression, Logistic; GLMM; Odds Ratio (OR) = 0.978, 95% CI 2-sided [0.702 to 1.361]
Statistical Analysis 3: Comparison: Intervention Arm vs Usual Care Arm; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.863, Regression, Logistic; GLMM; Odds Ratio (OR) = 0.961, 95% CI 2-sided [0.613 to 1.507]
Statistical Analysis 4: Comparison: Intervention Arm vs Usual Care Arm; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.963, Regression, Logistic; GLMM; Odds Ratio (OR) = 1.011, 95% CI 2-sided [0.636 to 1.607]

3. Other Pre Specified Outcome: COVID-19 Booster Vaccination
Description: Receipt of booster requires the Veteran needs to have completed the primary series of the COVID-19 vaccination.
Time Frame: 1 Year
Population: Veterans with at least one primary care visit and have completed the primary series either before or with enough time in the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 116319 | 143669
Participants | 56408 | 63909
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; No power calculation for this exploratory outcome. Null hypothesis is that both arms will have equal uptake rates of the COVID-19 Booster vaccination during the study period; Test type: Superiority; p = 0.395, Regression, Logistic — Threshold: P < 0.05; not adjusted for multiple comparisons; Generalized linear mixed modeling adjusted for baseline covariates and hierarchical levels for randomization units and clinics within them; Odds Ratio (OR) = 1.191, 95% CI 2-sided [0.796 to 1.781] — Odds ratio in favor of intervention arm (MI) has values higher than 1

4. Other Pre Specified Outcome: Receipt of Flu Vaccine
Description: Receipt of Flu Vaccine during study period.
Time Frame: 1 Year
Population: Veteran had to have at least one primary care visit during the study for primary analysis of this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 148291 | 190427
Participants | 76295 | 96561
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; Null hypothesis is that both study arms will have equal rates of flu vaccination uptake during the study period. No power calculation since this outcome is exploratory; Test type: Superiority; p = 0.119, Regression, Logistic — P-value was not adjusted for multiple comparisons and the p-value threshold was < 0.05; Generalized linear mixed model adjusting for baseline covariates and flu vaccine in prior year, with hierarchical random effects for ran. unit/site; Odds Ratio (OR) = 1.128, 95% CI 2-sided [0.97 to 1.311] — Odds ratio in favor of novel intervention arm has values higher than 1

ADVERSE EVENTS:
Time Frame: 1 Year of follow up
Arm/Group | Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/148291 | 0/190427
Serious Adverse Events (participants affected / at risk) | 0/148291 | 0/190427
Other Adverse Events (participants affected / at risk) | 0/148291 | 0/190427

LIMITATIONS AND CAVEATS:
Primary limitations were immunization ascertainment outside VHA. We supplemented using Medicare claims and state immunization registries, though neither covered the full period. VHA began querying state registries shortly before final data lock, with possible bias toward Veterans receiving more services. See SAP for details.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT05027464/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT05027464/SAP_002.pdf
  • Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT05027464/ICF_000.pdf